CLINICAL TRIAL: NCT03763721
Title: The ADVISE Study: Advanced Visualization In Corneal Surgery Evaluation Intra-operative Optical Coherence Tomography in Posterior Lamellar Keratoplasty
Brief Title: The ADVISE Study: Advanced Visualization In Corneal Surgery Evaluation
Acronym: ADVISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Maastricht University Medical Center (Other); Universitaire Ziekenhuizen KU Leuven (Other); Carl Zeiss Surgical GmbH (Industry)
Responsible Party: Principal Investigator, Robert P.L. Wisse, MD PhD, academic staff member, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL64392.041.17
Record Dates: First submitted 2018-11-15; First posted 2018-12-04 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Fuchs Dystrophy; Endothelial Corneal Dystrophy; Bullous Keratopathy; Vision Disorders
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal endothelial dystrophy type 2; Vision Disorders

STUDY DESIGN:
Intervention Model Description: The design of the study is a prospective, international, multicenter, non-inferiority, randomized controlled interventional clinical trial to compare the outcomes after posterior lamellar surgery with an iOCT optimized surgical protocol, and current practice, where the eye is over-pressurized for a set period of time. These groups will be labelled iOCT optimized protocol (iOCT-p) and current practice protocol (CP-p). Eligible patients will be assigned to either one of the groups. The study will be conducted simultaneously at the University Medical Center Utrecht (UMCU), Maastricht University Medical Center (MUMC) and the University Hospitals Leuven (UZL, Belgium). The inclusion, preoperative and postoperative measurements and questionnaires will take place at the Ophthalmology department of the site were the surgery was conducted. The research activities will be coordinated by the UMCU.
Who Masked: Participant
Masking Description: The patient will be blinded in the study, to prevent detection bias in filling out the questionnaires
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iOCT optimized protocol (iOCT-p) (Experimental): In the iOCT optimized protocol (iOCT-p) group, graft apposition will be assessed with special detail for graft orientation, interface fluid, and any peripheral folds as described by Xu et al. Potential tissue manipulations will be therefore based on the iOCT image. Apposition of the graft will be obtained using a complete filling of the anterior chamber with 20% sulphur hexafluoride (SF6) endotamponade for 1-2 minutes, whilst the OCT image is assessed and any graft manipulation can be performed if deemed necessary. After this period, the gas is partly exchanged for BSS (Balanced Salt Solution, Alcon) to achieve a bubble with a diameter of approximately the same size of the graft (i.e. 8.5mm)
  Interventions: Device: intraoperative optical coherence tomography (iOCT)
- current practice protocol (CP-p) (Active Comparator): In the current practice protocol (CP-p), graft apposition will be obtained using a complete and pressurized (approx. 65mmHg) filling of the anterior chamber with 20% SF6, for 8 minutes. Tissue manipulations, such as corneal swiping, will be performed as deemed necessary by the surgeon, based on the en face view from the conventional microscope image. The intraocular pressure is normalized by exchanging the SF6 gas for BSS, to achieve a gas bubble approximately the size of the graft (i.e 8.5mm). Now, the graft apposition is assessed using iOCT, to ensure all trial patients eventually undergo advanced iOCT imaging. Should this iOCT image reveal improper graft adherence or any other irregularity, the surgeon will perform additional manipulations or interventions as deemed necessary
  Interventions: Device: intraoperative optical coherence tomography (iOCT)

INTERVENTIONS:
Device: intraoperative optical coherence tomography (iOCT) — The OCT technology is fully integrated in a conventional ophthalmic surgical microscope (Zeiss LUMERA 700 platform). The OCT consists of A-scans (length/thickness) and B-scans (X-Y plane) to create the three dimensional image. Alternatively C-scans (3D cube scans) are available. All scans are non-invasive. The surgeon can continue surgery whilst using the iOCT and view a live image projected in the binocular or on the external screen and the video stream can be recorded as well.
  The iOCT features are controlled using the foot paddle and the images are recorded on device. Investigations will be performed in a standardized matter: iOCT imagery and cube-scans after graft insertion, air injection, and the end of surgery.

SUMMARY:
Rationale: Intra-operative optical coherence tomography (iOCT) is a new technology that incorporates advanced imaging techniques in the ophthalmic operating theatre. This allows surgeons to visualize tissues in a way previously impossible We conceptualized an iOCT-guided surgical protocol for the treatment of endothelial cell dysfunction, that refrains from the current practice of over-pressurizing the eye at the end of surgery.

Objective: The aim of this study is to assess the clinical value of intraoperative OCT (iOCT) for Descemet Membrane Endothelial Keratoplasty (DMEK) by comparing an iOCT-optimized surgical protocol with current practice, where the eye is over-pressurized for a set period of time, in terms of surgical efficiency, clinical outcomes, and adverse events.

Study design: International multicentre non-inferiority randomized clinical trial Study population: Patients scheduled for posterior lamellar corneal surgery for endothelial cell dysfunction above the age of 18 years.

Intervention: Both groups will undergo Descemet Membrane Endothelial Keratoplasty. Patients will be randomized for either the iOCT optimized surgical protocol or current standard surgical protocol using 8 minutes of overpressure to facilitate graft adherence. Both groups will be evaluated with iOCT at the end of surgery.

Main study parameters/endpoints:

The main study parameter is the rate of adverse events (particularly graft dislocations). Secondary parameters/endpoints are surgical time, the recovery of visual acuity and endothelial graft quality at 3 and 6 months follow-up, and a detailed evaluation of the extent/duration of surgical tissue manipulations.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The use of iOCT during surgery does not entail additional risk to the patient. Participants to this study will adhere to the standard of care after corneal transplant surgery. In addition, they will receive study specific measurements and questionnaires. The additional measurements and questionnaires will be combined with regular follow up moments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Irreversible corneal decompensation caused by Fuchs corneal endothelial dystrophy or pseudophakic bullous keratopathy
* Eligible for posterior lamellar keratoplasty, specifically Descemet Membrane Endothelial Keratoplasty (DMEK)

Exclusion Criteria:

* Any ocular co-morbidity other than cataract, mild dry eye disease, ocular hypertension, simple primary open angle glaucoma, and mild age-related macular degeneration
* Prior corneal transplant surgery
* Human leukocyte antigen (HLA) matched keratoplasty
* Any disability that will interfere with performing or understanding the procedures and questionnaire fulfilment except if it is temporary of nature.
* Combined phaco-emulsification-DMEK surgery (triple procedure)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
rate of the most relevant post-operative surgical complications | within 6 weeks post-operatively
  the number of patients that develop adverse events relating to lamellar corneal surgery, specifically graft detachments that necessitate a surgical intervention, early graft failures that lead to intractable corneal edema, or induced iatrogenic acute glaucoma

SECONDARY OUTCOMES:
Surgical time | during surgery
  times are recorded at entry of the OR, start time of the surgery, actual first incision, timepoint for injection of gas, duration of gas, closing time and departure time of the OR. Out of these both skin-to-skin and overall time in surgery can be calculated (i.e. gross/net)
Best-corrected visual acuity | 3 and 6 months follow-up
  Visual acuity is assessed using an ETDRS (Early Treatment Diabetic Retinopathy Study Chart) visual acuity chart with a spectacle correction. Visual acuity measurement ranges from light perception, hand movements, finger counting, 0.05 till 1.0. (US equivalent 20/20)
Graft endothelial cell densities | 3 and 6 months follow-up
  The quality of the graft is based on the amount and viability of endothelial cells. These will be measured (number of cells/mm2, variation in size (variation coefficient), hexagonality-coefficient) with in vivo specular microscopy.
Surgical manipulations | during surgery
  the recorded videos will be reviewed and scored considering the amount of surgical manipulations, the duration of all steps of the procedure, and the use of iOCT. All according to a study specific standard operating procedure

CONTACTS AND LOCATIONS:
Locations (3):
- Universiteitsziekenhuis Leuven, Leuven, Belgium
- Netherlands (2):
  - Maastricht University Hospital, Maastricht
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muijzer MB, Delbeke H, Dickman MM, Nuijts RMMA, Noordmans HJ, Imhof SM, Wisse RPL. Outcomes of the advanced visualization in corneal surgery evaluation trial; a non-inferiority randomized control trial to evaluate the use of intraoperative OCT during Descemet membrane endothelial keratoplasty. Front Ophthalmol (Lausanne). 2023 Jan 11;2:1041778. doi: 10.3389/fopht.2022.1041778. eCollection 2022. PMID 38983542
- [Derived] Muijzer MB, Delbeke H, Dickman MM, Nuijts RMMA, Jimale H, van Luijk CM, Imhof SM, Wisse RPL. Video Grading of Descemet Membrane Endothelial Keratoplasty Surgery to Identify Surgeon Risk Factors for Graft Detachment and Rebubbling: A Post Hoc Observational Analysis of the Advanced Visualization In Corneal Surgery Evaluation Trial. Cornea. 2023 Sep 1;42(9):1074-1082. doi: 10.1097/ICO.0000000000003181. Epub 2022 Nov 21. PMID 36730371
- [Derived] Muijzer MB, Noordmans HJ, Delbeke H, Dickman MM, Nuijts RMMA, Dunker S, Imhof SM, Wisse RPL. Establishing a Biomarker for the Prediction of Short-Term Graft Detachment After Descemet Membrane Endothelial Keratoplasty. Cornea. 2023 Feb 1;42(2):204-210. doi: 10.1097/ICO.0000000000003006. Epub 2022 Feb 18. PMID 35184123